CLINICAL TRIAL: NCT07288346
Title: Effect of Predictive Model on Total Double-Balloon Enteroscopy Rate: a Randomized Controlled Trial
Brief Title: Effect of Predictive Model on Double-Balloon Enteroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Qilu Hospital of Shandong University (Qingdao) (Other); Dezhou People's Hospital (Other); Yantai Affiliated Hospital of Binzhou Medical University (Other); Zaozhuang Municipal Hospital (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of the Qilu Hospital Gastroenterology Department, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: QLCR20250630
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Double-balloon Enteroscopy
MeSH Terms: interventions — Predictive Learning Models

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Predictive model group (Experimental): Endoscopists will obtain the predictive model intervention.
  Interventions: Other: Predictive model
- Control group (No Intervention): Endoscopists will not obtain the predictive model intervention.

INTERVENTIONS:
Other: Predictive model — Endoscopists obtain the patient's predictive model scores before double-balloon enteroscopy.
  Arms: Predictive model group

SUMMARY:
The aim of this study is to assess the effect of predictive model on total enteroscopy rate in double-balloon enteroscopy.

DETAILED DESCRIPTION:
Double-balloon enteroscopy is a new and effective endoscopic technique used for the diagnosis and treatment of small intestinal diseases. Due to its deep intubation ability, it can achieve complete visualization of the small intestinal mucosa, that is, total enteroscopy. Theoretically, a higher total enteroscopy rate could be associated with a greater possibility of detecting positive lesions. However, a total enteroscopy is a challenging procedure for endoscopists. Endoscopists cannot accurately predict the operational difficulty of patients before the operation, which leads to the passivity of preoperative preparation and intraoperative strategy formulation.

Recently, the Department of Gastroenterology of Qilu Hospital of Shandong University has completed the development and external validation of the first double-balloon enteroscopy prediction model. A preoperative individualized assessment of the difficulty of total enteroscopy can be achieved using this model. Therefore, a multicenter randomized controlled study was designed to assess the performance of predictive model in double-balloon enteroscopy, including total enteroscopy rate, positive findings, procedural time, adverse events and other indicators.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged between 18 and 80 years who were planned to undergo an attempt at total enteroscopy for suspected small-bowel disease
2. CT scan of the abdomen was performed within two weeks before enteroscopy

Exclusion Criteria:

1. cases terminated upon the target lesion (strictures, masses, hemorrhagic or other lesions) and not the maximal insertion
2. poor quality of bowel preparation
3. high risk esophageal varices
4. the insertion route is not oral or anal because of changes in anatomical structure
5. unsuitable for general anesthesia
6. pregnant women
7. unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Total enteroscopy rate | 8 months
  Total enteroscopy rate was defined as the number of patients with complete visualization of the small bowel divided by the total number of patients.

SECONDARY OUTCOMES:
Diagnostic yield | 8 months
  Positive findings included vascular malformation, ulcer, polyp, diverticulum and others.
Procedural time | 8 months
  The total time of antegrade and retrograde insertions
Adverse events | 8 months
  Adverse reactions refer to bleeding, perforation, aspiration pneumonia, acute pancreatitis and other conditions related to double-balloon enteroscopy.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Dezhou People's Hospital, Dezhou, Shandong
  - Qilu Hospital of Shandong University (Qingdao), Qingdao, Shandong
  - Yantai Affiliated Hospital of Binzhou Medical University, Yantai, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shangdong